CLINICAL TRIAL: NCT02141984
Title: Post-Marketing Surveillance of Humira Injection in Korean JIA Patients Under the New-Drug Re-examination
Brief Title: Surveillance of Humira in Korean JIA Patients
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P14-362
Record Dates: First submitted 2014-05-16; First posted 2014-05-20 (Estimated); Results first posted 2017-06-23 (Actual); Last update posted 2017-06-23 (Actual); Status verified 2017-04

CONDITIONS: Polyarticular Juvenile Idiopathic Arthritis
Keywords: Korean regulatory required Postmarketing Surveillance
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with Polyarticular JIA or ERA: Patients with polyarticular juvenile idiopathic arthritis (JIA) or enthesitis-related arthritis (ERA)

SUMMARY:
Approximately 600 pediatric patients prescribed Humira Injection in usual practice according to the approved Korean product label will be registered into this observational study. Baseline data will be obtained at enrollment including demographics, underlying diseases and complications especially in regard to purified protein derivative (PPD) skin test, and chest X-ray. At routine visits for Humira Injection administration, which will occur according to usual medical practice, concomitant medication information and adverse events information will be collected for up to 70 days after the last administration of Humira.

ELIGIBILITY:
Inclusion Criteria:

* Patients from 2 years of age who were diagnosed with polyarticular juvenile idiopathic arthritis (JIA) or patients from 6 years of age who were diagnosed with enthesitis-related arthritis (ERA).
* Polyarticular juvenile idiopathic arthritis (JIA) patients for whom the response to previous disease-modifying anti rheumatic drug therapy has been inadequate
* Patients who give written authorization form to use their personal and health data from legal parents or representative.
* Physician will refer to the product market authorization (label) for inclusion criteria.

Exclusion Criteria:

* Patients with known hypersensitivity to Humira or any of its excipients.
* Patients who is participating on other clinical trials.
* Physician will refer to the product market authorization (label) for exclusion criteria.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: General hospital
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2014-05; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eunjung Gu, MS, Study Director — AbbVie korea

REFERENCES:
- See also: Related Info — http://rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 600 participants were expected to enroll in the study; however, due to low prevalence of JIA and ERA, only 28 participants were enrolled.
Period: Overall Study
Arm/Group | Patients With Polyarticular JIA or ERA
Started | 28
Completed | 26
Not Completed | 2
Not completed — Lack of Efficacy | 2

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Polyarticular JIA or ERA
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.68 (5.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. The investigator assessed the relationship of each event to the use of study drug as either related, possible, probably not, not related, or unassessable. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the subject and may require medical or surgical intervention to prevent any of the outcomes listed above.
Time Frame: Adverse Events (AEs) were collected from informed consent to within 70 days following the last scheduled administration of Humira (up to 22 weeks)
Population: Safety analysis set: All participants who received at least one administration of Humira during the study (after informed consent or first administration of Humira) and for 70 days following the last scheduled administration of Humira.
Measure: Number; unit: participants
Arm/Group | Patients With Polyarticular JIA or ERA
Number analyzed (Participants) | 28
participants
  Any AE | 6
  Unexpected AE | 1
  Any SAE | 1

2. Secondary Outcome: Changes in Active Joint Count From Baseline and 12 Weeks Post-Treatment
Description: Active Joint Count will be assessed and collected by participating investigators in routine medical practice. Sixty-eight joints were assessed by physical examination. Active joints are defined as joints with positive results for tenderness, swelling, pain on passive motion, or limitation of passive motion. Higher scores represent higher disease activity.
Time Frame: From the first administration (Day 1) to approximately 12 weeks (±4 weeks)
Population: Effectiveness analysis set: All participants who have been administered Humira for not less than 12 (± 4) weeks or more and for whom effectiveness evaluation parameters have been recorded including active joint count as well as Physician global assessment and Parent's global assessment at baseline and 12 weeks.
Measure: Mean (Standard Deviation); unit: active joint
Arm/Group | Patients With Polyarticular JIA or ERA
Number analyzed (Participants) | 19
active joint | -6.05 (6.65)

3. Secondary Outcome: Physician's Global Assessment of the Disease
Description: The Physician's global assessment of the disease assessment was evaluated as 'Improved,' 'Not changed,' 'Aggravated,' or 'Not assessable.'
Time Frame: From the first administration (Day 1) to approximately 12 weeks (±4 weeks)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Patients With Polyarticular JIA or ERA
Number analyzed (Participants) | 19
participants
  Improved | 18
  Not changed | 1
  Aggravated | 0
  Not assessable | 0

4. Secondary Outcome: Parent's Global Assessment for Effectiveness
Description: Parent's global assessment for effectiveness was evaluated as 'Improved,' 'Not changed,' 'Aggravated,' or 'Not assessable.'
Time Frame: From the first administration (Day 1) to approximately 12 weeks (±4 weeks)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Polyarticular JIA or ERA
Number analyzed (Participants) | 19
Participants
  Improved | 19
  Not changed | 0
  Aggravated | 0
  Not assessable | 0

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from first dose of study drug until 70 days after the last dose of study drug (up to 22 weeks); SAEs were collected from the time informed consent was obtained (22 weeks).
Arm/Group | Patients With Polyarticular JIA or ERA
Serious Adverse Events (participants affected / at risk) | 1/28
Other Adverse Events (participants affected / at risk) | 6/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients With Polyarticular JIA or ERA (N=28)
Erythema (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients With Polyarticular JIA or ERA (N=28)
Influenza (Infections and infestations) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Pyrexia (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.